CLINICAL TRIAL: NCT05137275
Title: Dose Escalation and Extension Study to Evaluate the Safety, Tolerability, and Initial Efficacy of Anti-5T4 CAR-raNK Cell Therapy in Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of Anti-5T4 CAR-raNK Cell Therapy in Locally Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Collaborators: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jin Li, Director, Shanghai East Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IBR854-03
Record Dates: First submitted 2021-11-11; First posted 2021-11-30 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-5T4 CAR-raNK Cells (Experimental)
  Interventions: Biological: Anti-5T4 CAR-raNK Cells

INTERVENTIONS:
Biological: Anti-5T4 CAR-raNK Cells — In the 3+3 dose escalation study, the minimum initial dose is 3.0×10^9 cells and then escalate to 6.0× 10^9 and 9.0× 10^9 cells. Every 21 days is one cycle, and intravenous infusion is performed on day 1 and day 3\8 of each cycle. In dose extension study, the initial dose will be determined by RP2D determined by the results of dose escalation study, and the other intervention methods are consistent.

SUMMARY:
This study is a multicenter, open-label, investigator-initiated trial (IIT), divided into dose escalation (Part A) and dose extension (Part B) phases to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacokinetics (PD) and initial efficacy of conjugated antibody redirecting ready-to-use allogeneic NK (CAR-raNK) cells that target trophoblast glycoprotein (5T4) in patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Part A is a dose escalation study to evaluate maximum toxic dose (MTD) and/or recommended phase II dose (RP2D) which adopts the 3+3 dose escalation design protocol. The dose is respectively 3.0×10^9 live cells, 6.0×10^9 live cells and 9.0×10^9 live cells (if the safety of dose group with 9.0×10^9 live cells is still good, the Safety Monitoring Committee (SMC) will co-decide whether to continue the dose escalation and the specific dose based on the obtained data on safety, efficacy, and PK). The 3.0×10^9 live cell dose group is given on days 1 and 3 of each cycle (21 days), and the follow-up dose group is given on days 1 and 8 of each cycle (21 days).3-6 subjects will be enrolled at every dose level. The first and second subjects in the same group shall be enrolled at an interval of at least 7 days, for the purpose of ensuring their safety. Only when the dose-limiting toxicity (DLT) of all subjects in the previous dose group was observed can the enrollment of the next dose group get started.

Part B is the dose extension study. After recommended phase II dose (RP2D) is determined in Part A, the SMC will discuss whether to conduct the Part B study. This stage will be carried out in different tumor types with high expression of 5T4 antigen, and 6 to 10 subjects will be enrolled in each tumor type, and all subjects will receive anti-5T4 CAR-raNK cell therapy at RP2D level. Every 21 days is one cycle, and the administration is performed on day 1 and day 8 of each cycle.

ELIGIBILITY:
Inclusion criteria:

1. Subjects volunteer to participate in this clinical study, are fully aware of the study and have signed the Informed Consent Form (ICF). Subjects are willing to follow and able to complete all trial procedures.
2. Age: adult at the age of 18-80 (both inclusive), female or male. Patients with advanced malignant solid tumors, histologically or cytologically confirmed, who had failed standard therapy, or had no standard therapy, or were not eligible for standard therapy at this stage; Part B: Patients with specific primary tumor types, including:

   * Cohort 1: Non-small cell lung cancer with disease progression or intolerance after at least two systemic therapies; For patients with known epidermal growth factor receptor (EGFR)-sensitive mutations, anaplastic lymphoma kinase (ALK) gene fusion, or other driver gene positivity, progression must be followed by appropriate targeted therapy.
   * Cohort 2: Breast cancer, negative for progesterone receptor (PR), estrogen receptor (ER), and human epidermal growth factor receptor-2 (HER2), treated with at least one systemic chemotherapy agent.
   * Cohort 3: Colorectal cancer with disease progression or intolerance after at least two systemic therapies.
   * Cohort 4: Mesothelioma with disease progression or intolerance after at least two systemic therapies.
   * Cohort 5: Other tumors with high expression of antigen 5T4.
3. Eastern Cooperative Oncology Group (ECOG) score ≤1 and expected survival time > 3 months.
4. (Part A) According to RECIST v1.1, there is at least one assessable tumor lesion; (Part B) According to RECIST v1.1, there is at least one measurable tumor lesion (a lesion within the field of previous radiation cannot be targeted unless there is radiographic evidence of progression or persistence after 3 months of radiation).
5. Organ function during screening should meet the following criteria:
6. Hematologic system (no blood transfusion or hematopoietic stimulator treatment within 14 days)

   * Absolute neutrophil count (ANC) ≥1.5×109/L
   * Platelet (PLT) ≥75×109/L
   * Hemoglobin (Hb) ≥85g/L
   * Hepatic function
   * Total bilirubin (TBIL) ≤1.5×ULN
   * Alanine aminotransferase (ALT) ≤3×ULN;
   * Patients with liver metastasis or liver cancer: ≤5×ULN
   * Aspartate aminotransferase (AST) ≤3×ULN;
   * Patients with liver metastasis or liver cancer: ≤5×ULN Renal function
   * Creatinine (Cr) ≤1.5× ULN
   * Creatinine clearance (Ccr) (to be calculated only when Cr > 1.5× ULN) > -50ml/min/1.73m2 (Cockcroft-Gault formula) Coagulation function
   * Activated partial thrombin time (APTT) ≤1.5×ULN
   * International normalized ratio (INR) ≤1.5×ULN
7. Subjects of reproductive age and their partners should agree to have no family planning and to use effective contraceptive methods (hormonal or barrier methods or abstinence, etc.) for 6 months from signing the ICF until the last dose of the study drug is administered; women of reproductive age must have a negative serological pregnancy test 7 days prior to their first use of the study drug.

Exclusion Criteria:

1. Have received systemic antitumor therapy, including chemotherapy, immunotherapy, and radical radiotherapy, within 4 weeks prior to their first use of the study drug. The following special cases should be assessed separately:

   * The time of the last treatment of nitrosourea or mitomycin C is less than 6 weeks before the first use of the study drug;
   * The time of last treatment of fluorouracil and small-molecule targeted drugs is less than 2 weeks or 5 half-lives of the drug (whichever was longer) after the first use of the study drug;
   * The time of the last treatment of the traditional Chinese medicine with anti-tumor indications was less than 2 weeks after the first use of the study drug.
2. Have participated in other clinical trials and received any unmarketedinvestigational drug or treatment within 4 weeks prior to first use of the study drug.
3. Any prior adoptive cellular immunotherapy.
4. Have undergone major organ surgery (excluding needle biopsy) or had significant trauma within 4 weeks prior to their first use of the study drug, or required elective surgery during the study period.
5. Have received systemic glucocorticoids (prednisone> 10 mg/ day or an equivalent dose of another drug of the same class) or other immunosuppressants within 14 days prior to initial use of the study drug. The exceptions are: local, ocular, intraarticular, intranasal, and inhaled glucocorticoids; short-term use of glucocorticoids for prophylaxis (e.g., to prevent contrast allergy).
6. Have received live, attenuated, adenovirus, or messenger ribonucleic acid (mRNA) vaccines within 4 weeks prior to initial use of the study drug, or plan to receive these vaccines during the study period.
7. Have used immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc., within 14 days prior to their first use of study drugs.
8. Patients with active infection who currently require intravenous anti-infective therapy.
9. Active hepatitis b (HBsAg positive and hepatitis b virus (HBV) DNA
10. Patients with a known history of human immunodeficiency virus (HIV) infection, or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
11. Have active autoimmune diseases or have had autoimmune diseases that are likely to recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, psoriasis, etc.). Except in the following cases: type 1 diabetes that was well controlled with hormone replacement therapy, hypothyroidism, skin conditions that did not require systemic therapy (e.g., vitiligo), and other conditions that were well controlled and that the investigator determined were less likely to recur (e.g., childhood asthma in remission).
12. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    * There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia, and Ⅱ-Ⅲ degree atrioventricular block, which need clinical intervention;
    * The mean QT interval (QTcF) corrected by Fridericia method was > 480ms;
    * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurring within 6 months before the first administration;
    * Patients with heart failure or left ventricular ejection fraction (LVEF) < 50% in the New York Heart Association (NYHA) classification ≥II;
    * Hypertension beyond clinical control.
13. Previous or current interstitial lung disease (except local interstitial pneumonia induced by radiotherapy).
14. Adverse effects of previous antineoplastic therapy have not returned to CTCAE grade 5.0 ≤1 (except for toxicity that the investigator determined to be of no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy).
15. Cerebral parenchymal metastasis or meningeal metastasis with clinical symptoms were deemed unsuitable for inclusion by the investigator.
16. Had received immunotherapy and developed grade ≥3 immune-related adverse events (irAE).
17. The third interstitial effusion, which could not be controlled clinically, was judged by the investigator to be unsuitable for inclusion.
18. (Extension phase) had other malignant tumors in the past 5 years, excluding skin basal cell carcinoma, ductal carcinoma in situ and cervical carcinoma in situ with a radical surgery.
19. Pregnant or lactating women.
20. Have a history of alcohol or drug abuse.
21. Mental disorder or poor compliance.
22. The investigator considered that the subjects had a history of other serious systemic diseases or other reasons that made them unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of dose limiting toxicity (DLTs) | From day1 to day 21
  To evaluate the safety, tolerability, and determine the RP2D of Anti-5T4 CAR-raNK Cells
Part A: Number of Adverse Events (AEs) | From day 1 to day 90 after the last dose
  To evaluate the safety of Anti-5T4 CAR-raNK Cells
Part B: Objective response rate (ORR) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of Anti-5T4 CAR-raNK Cells
Part B: Disease control rate (DCR) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of Anti-5T4 CAR-raNK Cells
Part B: Duration of remission (DOR) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of Anti-5T4 CAR-raNK Cells
Part B: Progression-free survival (PFS) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of Anti-5T4 CAR-raNK Cells
Part B: Overall survival (OS) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of Anti-5T4 CAR-raNK Cells

SECONDARY OUTCOMES:
The number of CAR-raNK cells | From day1 to day 21
  Blood samples will be collected at specified time points to detect the number of CAR raNK cells in peripheral blood
Cytokine release | From day1 to day 21
  Blood samples will be collected at specified time points to detect serum Blood samples will be collected at specified time points to detect the cytokine (IL-1β, IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α) concentration
Lymphocyte subtype | From day1 to day 21
  Blood samples will be collected at specified time points to analyze the lymphocyte subtypes (CD3, CD4, CD8, CD19, CD56).
Anti-CAR antibodies | From day1 to day 21
  Blood samples will be collected at specified time points to detect anti-CAR(anti-5T4 mAb) antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gras Navarro A, Bjorklund AT, Chekenya M. Therapeutic potential and challenges of natural killer cells in treatment of solid tumors. Front Immunol. 2015 Apr 29;6:202. doi: 10.3389/fimmu.2015.00202. eCollection 2015. PMID 25972872
- [Background] Franks SE, Wolfson B, Hodge JW. Natural Born Killers: NK Cells in Cancer Therapy. Cancers (Basel). 2020 Jul 31;12(8):2131. doi: 10.3390/cancers12082131. PMID 32751977
- [Background] Griffiths RW, Gilham DE, Dangoor A, Ramani V, Clarke NW, Stern PL, Hawkins RE. Expression of the 5T4 oncofoetal antigen in renal cell carcinoma: a potential target for T-cell-based immunotherapy. Br J Cancer. 2005 Sep 19;93(6):670-7. doi: 10.1038/sj.bjc.6602776. PMID 16222313
- [Background] Shaw DM, Embleton MJ, Westwater C, Ryan MG, Myers KA, Kingsman SM, Carroll MW, Stern PL. Isolation of a high affinity scFv from a monoclonal antibody recognising the oncofoetal antigen 5T4. Biochim Biophys Acta. 2000 Dec 15;1524(2-3):238-46. doi: 10.1016/s0304-4165(00)00165-3. PMID 11113573
- [Background] Redchenko I, Harrop R, Ryan MG, Hawkins RE, Carroll MW. Identification of a major histocompatibility complex class I-restricted T-cell epitope in the tumour-associated antigen, 5T4. Immunology. 2006 May;118(1):50-7. doi: 10.1111/j.1365-2567.2006.02338.x. PMID 16630022
- [Background] Stern PL, Harrop R. 5T4 oncofoetal antigen: an attractive target for immune intervention in cancer. Cancer Immunol Immunother. 2017 Apr;66(4):415-426. doi: 10.1007/s00262-016-1917-3. Epub 2016 Oct 18. PMID 27757559
- [Background] Liu E, Marin D, Banerjee P, Macapinlac HA, Thompson P, Basar R, Nassif Kerbauy L, Overman B, Thall P, Kaplan M, Nandivada V, Kaur I, Nunez Cortes A, Cao K, Daher M, Hosing C, Cohen EN, Kebriaei P, Mehta R, Neelapu S, Nieto Y, Wang M, Wierda W, Keating M, Champlin R, Shpall EJ, Rezvani K. Use of CAR-Transduced Natural Killer Cells in CD19-Positive Lymphoid Tumors. N Engl J Med. 2020 Feb 6;382(6):545-553. doi: 10.1056/NEJMoa1910607. PMID 32023374
- [Background] Xia H, Wang Y, Sun HL, Gao LY, Cao Y, Zaongo SD, Zeng RN, Wu H, Zhang MJ, Ma P. Safety and efficacy of allogeneic natural killer cell immunotherapy on human immunodeficiency virus type 1 immunological non-responders: a brief report. Chin Med J (Engl). 2020 Dec 5;133(23):2803-2807. doi: 10.1097/CM9.0000000000001189. PMID 33273328
- [Background] Nagai K, Harada Y, Harada H, Yanagihara K, Yonemitsu Y, Miyazaki Y. Highly Activated Ex Vivo-expanded Natural Killer Cells in Patients With Solid Tumors in a Phase I/IIa Clinical Study. Anticancer Res. 2020 Oct;40(10):5687-5700. doi: 10.21873/anticanres.14583. PMID 32988894